CLINICAL TRIAL: NCT02317653
Title: Mom2Baby Pilot: Understanding the Influence of Pregnancy on Breast Milk
Brief Title: Understanding the Influence of Pregnancy on Breast Milk
Acronym: Mom2Baby Pilot
Status: Completed | Type: Observational
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Henry J. Nuss, Ph.D., Assistant Professor, Louisiana State University Health Sciences Center in New Orleans
Other Study IDs: PBRC2014-049
Record Dates: First submitted 2014-12-08; First posted 2014-12-16 (Estimated); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Pregnancy; Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Maternal Blood Collection: approximately 60 mL of blood will be collected over 2 timepoints
  Breast Milk Collection: approximately 50-100 mL of breast milk will be collected at 1 timepoint
  Infant Stool Collection: 1 fresh infant stool sample will be collected at 1 timepoint
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Overweight/Obese: Archive blood, archive breast milk, and clinical assessment data from 15 participants who were considered overweight or obese at enrollment in the Expecting Success study conducted at Pennington Biomedical Research Center (NCT01610752) will be used to represent the overweight and obese sample for study investigations.
- Normal Weight: Up to 20 pregnant women who were considered normal weight (18.5 ≤ BMI ≤ 24.9 kg/m2) prior to pregnancy will be enrolled in the study.

SUMMARY:
The purpose of this study is to identify the influences of pregnancy on breast milk and the effects of these on the health of babies during the first 2 months of life. The investigators hypothesize that overweight and obese mothers will have lower serum n-3 to n-6 PUFA ratios during pregnancy and postpartum than normal weight mothers and will be positively correlated with TNF-α, IL-1β, resistin, and negatively correlated ghrelin levels both in serum and in breast milk in postpartum.

DETAILED DESCRIPTION:
The Mom2Baby Pilot study will last about 4 months. Up to 20 pregnant women who were considered normal weight prior to pregnancy will be enrolled in the study. The infants born to these pregnant women will also be enrolled after birth. Archive blood, archive breast milk, and clinical assessment data from up to 20 participants who were considered overweight or obese at enrollment in the Expecting Success study conducted at Pennington Biomedical Research Center (NCT01610752) may be used to test the primary hypothesis as well as additional hypotheses.

We will measure levels of LC-PUFAS, pro-inflammatory biomarkers, and regulatory hormones (resistin, ghrelin) in serum (35,0-36,6 weeks gestation and 4,0-7,6 weeks postpartum) and breast milk (4,0-7,6 weeks postpartum) in normal weight (n=20) and overweight and obese (n=20) mothers. Blood serum and plasma and breast milk levels of these measures will be compared from pregnancy to postpartum within and between normal weight and overweight and obese women. Additional maternal procedures including questionnaires, anthropometrics, body composition measurements, energy intake measurement, and physical activity measurement will be investigated at 35,0-36,6 weeks gestation and 4,0-7,6 weeks postpartum. Infant procedures including anthropometrics, body composition measurements, stool collection, and energy intake measurement will be investigated at 0,1-0,6 weeks and 4,0-7,6 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Pregnant (prior to 36 weeks gestation) with singleton viable pregnancy
* Not diagnosed with gestational diabetes in the 2nd trimester of current pregnancy as determined by 2nd trimester oral glucose tolerance test
* 18-40 years of age
* Normal weight (18.5 ≤ BMI ≤ 24.9 kg/ m2) prior to pregnancy
* English speaking
* Willing to complete up to 3 clinic visits at Pennington Biomedical Research Center
* Willing to enroll infant in the study after infant is delivered
* Intend to breastfeed or provide breast milk to infant until the infant is at least 2 months of age
* Willing for study staff to contact the primary care doctor who is providing prenatal care for the current pregnancy and to obtain information from the prenatal medical records, the labor and delivery records and the medical records of the infant at birth

Exclusion Criteria:

* Recent history of or currently smoking
* Recent history of or current alcohol or drug abuse
* Not willing to complete up to 3 clinic visits at Pennington Biomedical Research Center
* Not willing to enroll infant in the study after infant is delivered
* Not planning on breastfeeding or providing breast milk to infant prior to 2 months of age
* Plans to move out of the study area within the study period
* Not willing to avoid pregnancy for 2 months following delivery
* Prior or planned (within 1 year of expected delivery) bariatric surgery
* Enrollment in this study in a previous pregnancy
* Known fetal anomaly in current pregnancy
* History of preterm birth
* Planned termination or adoption of infant from current pregnancy
* History of 3 or more consecutive first trimester miscarriages
* Hypertensive (SBP>160 mmHg & DBP >110 mmHg)
* Diabetic diagnosis prior to pregnancy
* History or current psychotic disorder, major depressive episode, bipolar disorder, or eating disorder
* Diagnosis of HIV or AIDS
* Diagnosis of severe anemia (Hb<8g/dL and/or Hct <24%)
* Current use of one or more of the following medications: Metformin, Systemic steroids, Antipsychotic agents (e.g., Abilify, Haldol, Risperdal, Seroquel, Zyprexa), Anti-seizure medications or mood stabilizers that would be expected to have a significant impact on body weight (e.g., Depakote, Lamictal, Lithium, Neurontin, Tegretol, Topamax, Keppra), Medications for ADHD including amphetamines and methylphenidate.
* Continued use of weight loss medication including OTC and dietary supplements for weight loss (e.g.,Adipex, Suprenza, Tenuate, Xenical, Alli, conjugated linoleic acid, Hoodia, Green tea extract, Guar gum, HydroxyCut, Sensa, Corti-slim, Chromium, chitosan, Bitter orange)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Up to 20 pregnant women who were considered normal weight (18.5 ≤ BMI ≤ 24.9 kg/m2) prior to pregnancy will be enrolled in the study.
  Archive blood, archive breast milk, and clinical assessment data from 15 participants who were considered overweight and obese at enrollment in the Expecting Success study conducted at Pennington Biomedical Research Center (NCT01610752) will be used to represent the overweight and obese sample.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
serum levels of n-3 to n-6 PUFA ratios during pregnancy will be compared to inflammatory markers and regulatory markers in blood and breast milk in both groups | 1-2 months postpartum

SECONDARY OUTCOMES:
energy intake and diet quality assessed compositely with the Remote Food Photography Method developed at Pennington Biomedical during pregnancy will be compared to energy intake and diet quality in postpartum in both groups. | 1-2 months postpartum

OTHER OUTCOMES:
n-3 and n-6 PUFA levels and inflammatory markers in mother's blood and breast milk will be assessed to test correlations to infants' body composition | 1-2 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Henry Nuss, Ph.D., Principal Investigator — Louisiana State University Health Sciences Center in New Orleans
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States